CLINICAL TRIAL: NCT02297412
Title: Pilot Clinical Trial Evaluating the Utility of Minocycline as an Agent to Decrease Chemotherapy-Induced Peripheral Neuropathy (CIPN) and Paclitaxel-Induced Acute Pain Syndrome (P-APS): A Randomized Placebo-Controlled, Double Blind Trial
Brief Title: Minocycline Hydrochloride in Reducing Chemotherapy-Induced Peripheral Neuropathy and Acute Pain in Patients With Breast Cancer Undergoing Treatment With Paclitaxel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RU221408I; NCI-2016-01592 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RU221408I (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2014-11-14; First posted 2014-11-21 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Acute Pain; Breast Carcinoma; Peripheral Neuropathy
MeSH Terms: conditions — Acute Pain; Breast Neoplasms; Peripheral Nervous System Diseases | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (minocycline hydrochloride) (Experimental): Patients receive minocycline hydrochloride PO BID on days 1-7. Treatment repeats every 7 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Minocycline Hydrochloride; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (placebo) (Placebo Comparator): Patients receive a placebo PO BID on days 1-7. Treatment repeats every 7 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Placebo; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Minocycline Hydrochloride — Given PO
  Other Names: Dynacin; Minocin; Minomax; Minomycin; Tri-minocycline; Vectrin
  Arms: Arm I (minocycline hydrochloride)
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized pilot trial studies how well minocycline hydrochloride works in reducing chemotherapy-induced peripheral neuropathy and acute pain in patients with breast cancer undergoing treatment with paclitaxel. Drugs used in chemotherapy, such as paclitaxel, may cause damage to nerves that result in aches, pains, and tingling or numbness of fingers and toes. Minocycline hydrochloride may help lessen nerve damage from paclitaxel and improve the quality of life in breast cancer patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate whether minocycline hydrochloride (minocycline) can alleviate paclitaxel-induced peripheral neuropathy.

II. To estimate whether minocycline can alleviate paclitaxel acute pain syndrome (P-APS).

III. To examine the possible relative toxicities related to minocycline therapy in this study situation.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive minocycline hydrochloride orally (PO) twice daily (BID) on days 1-7. Treatment repeats every 7 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive a placebo PO BID on days 1-7. Treatment repeats every 7 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of the study, patients are followed up every month for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Ability to complete questionnaires by themselves or with assistance
* Planned paclitaxel at a dose of 80 mg/m2 IV given, in the adjuvant breast cancer (postoperative or neo-adjuvant) setting, every week for a planned course of 12 weeks without any other concurrent cytotoxic chemotherapy (trastuzumab and/or other antibody and/or small molecule treatment is allowed, except for PARP inhibitors)
* Life expectancy > 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Negative pregnancy test (serum or urine) done =< 7 days prior to registration, for women of childbearing potential only (determined per clinician discretion)

Exclusion Criteria:

* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Previous diagnosis of diabetic neuropathy or peripheral neuropathy from any cause
* History of allergic or other adverse reactions to minocycline
* Prior exposure to neurotoxic chemotherapy
* Diagnosis of fibromyalgia
* Current or planned use of methoxyflurane, oral contraceptives, isotretinoin, penicillin, or ergot alkaloids
* History of allergic or other adverse reactions to tetracycline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-11; Primary Completion 2016-07-08 (Actual); Study Completion 2016-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Loprinzi, Principal Investigator — Academic and Community Cancer Research United
Locations (12):
- United States (12):
  - PCR Oncology, Pismo Beach, California
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Women and Infants Hospital, Providence, Rhode Island
  - Marshfield Clinic, Marshfield, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Minocycline Hydrochloride) | Arm II (Placebo)
Started | 23 | 24
Completed | 22 | 23
Not Completed | 1 | 1
Not completed — Canceled | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Minocycline Hydrochloride) | Arm II (Placebo) | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (10.1) | 55.0 (11.8) | 54.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 23 | 45

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) Per Assessment (aAUCpa) of Average Pain (Item 3 on the Daily Post-Paclitaxel Questionnaire)
Description: Average Area Under the Curve (AUC) per assessment (aAUCpa) of average pain (item 3 on the Daily Post-Paclitaxel Questionnaire; "Please rate the same aches/pain by circling the ONE number that best describes your aches/pains on the AVERAGE in the last 24 hours.") over 12 weeks. Scores are reported on a 0-100 scale, where 100=better outcome quality of life (QOL). The aAUCpa is the average of each AUC between each sequential assessment from treatment-initiation to the week-12 assessment.
Time Frame: Up to 12 weeks
Population: Patients who completed the Daily Post-Paclitaxel Questionnaire item 3 over 12 weeks were included in this analysis.
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Arm I (Minocycline Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 20 | 20
scores on a scale | 96.0 [54.4 to 100.0] | 84.3 [46.5 to 99.7]
Statistical Analysis 1: Comparison: Arm I (Minocycline Hydrochloride) vs Arm II (Placebo); Test type: Superiority or Other; p = 0.0186, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Area Under the Curve (AUC) of EORTC CIPN20 Sensory Neuropathy Subscale
Description: Average Area Under the Curve per assessment (aAUCpa) of EORTC Chemotherapy-Induced Peripheral Neurophathy Module (EORTC QLQ-CIPN20) Sensory Neuropathy Subscale. The EORTC CIPN20 scoring algorithm was used for the sensory (items 31-36, 39, 40 and 48) subscale scores on a 0-100 scale, with higher scores represent fewer symptoms (better QOL). The aAUCpa for the subscale is calculated as the average of each AUC between each sequential assessment from treatment-initiation to the week-12 assessment. For example; for each patient and each subscale, the subscale values at treatment-initiation and assessment-1 are used to calculate an Area Under the Curve (AUC) for that assessment time-period. Then these AUCs for all available assessment time-periods up to week-12 are averaged to yield the aAUCpa per patient per subcale.
Time Frame: Up to course 12
Population: Patients who completed the EORTC Chemotherapy-Induced Peripheral Neurophathy Module Sensory Neuropathy Subscale items over 12 weeks were included in this analysis.
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Arm I (Minocycline Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 21 | 20
scores on a scale | 94.1 [58.7 to 100.0] | 89.4 [68.7 to 98.3]
Statistical Analysis 1: Comparison: Arm I (Minocycline Hydrochloride) vs Arm II (Placebo); Test type: Superiority or Other; p = 0.1146, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Area Under the Curve (AUC) Per Assessment (aAUCpa) of Fatigue (Item 10 on the Acute Pain Syndrome Summary Questionnaire)
Description: Area Under the Curve (AUC) Per Assessment (aAUCpa) of Fatigue (Item 10 on the Acute Pain Syndrome Summary Questionnaire); "Over the past week, did you experience fatigue?") over 12 weeks. Scores are reported on a 0-100 scale, where 100=better outcome quality of life (QOL). The aAUCpa is the average of each AUC between each sequential assessment from treatment-initiation to the week-12 assessment.
Time Frame: Baseline to up to 12 weeks
Population: Patients who completed the Acute Pain Syndrome Summary Questionnaire over 12 weeks are included in this analysis.
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Arm I (Minocycline Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 21 | 21
scores on a scale | 76.7 [30.8 to 90.0] | 59.0 [29.4 to 86.4]
Statistical Analysis 1: Comparison: Arm I (Minocycline Hydrochloride) vs Arm II (Placebo); Test type: Superiority or Other; p = 0.0243, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Description: The descriptions & grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting. Each CTCAE term in the current version is a unique representation of a specific event used for medical documentation & scientific analysis & is a single MedDRA Lowest Level Term (LLT).
Arm/Group | Arm I (Minocycline Hydrochloride) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 3/22 | 1/23
Other Adverse Events (participants affected / at risk) | 8/22 | 9/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Minocycline Hydrochloride) (N=22) | Arm II (Placebo) (N=23)
Lung infection (Infections and infestations) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Minocycline Hydrochloride) (N=22) | Arm II (Placebo) (N=23)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (3) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (3) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (10)
Dizziness (Nervous system disorders) | 1 (3) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (7)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No